CLINICAL TRIAL: NCT01775267
Title: ASSOCIATING LIVER PARTITION WITH PORTAL VEIN LIGATION FOR STAGED HEPATECTOMY (ALPPS) Versus Conventional Portal Vein Occlusion (PVO) for Resection of Liver Tumors Unresectable in One Step - a Randomized Controlled Trial
Brief Title: ALLPS VERSUS PVO Randomized Controlled Trial
Acronym: ALPPS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to safety concerns in both study arms
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USZ-ZH-VIS-ALPPS
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Liver Tumors Not Resectable in One Surgical Procedure
MeSH Terms: interventions — Ligation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALPPS (Experimental): Patients undergo Liver partition and portal vein ligation to induce hypertrophy of the future liver remnant
  Interventions: Procedure: Associating liver partition and portal vein ligation for staged hepatectomy
- PVO (Active Comparator): Patient undergo portal vein embolization or ligation
  Interventions: Procedure: Portal vein embolization or ligation

INTERVENTIONS:
Procedure: Associating liver partition and portal vein ligation for staged hepatectomy
  Arms: ALPPS
Procedure: Portal vein embolization or ligation
  Arms: PVO

SUMMARY:
This randomized phase II trial compares how well associating liver partition with portal vein ligation for staged hepatectomy (ALPPS) or portal vein occlusion (PVO) works in treating patients with liver cancer. Both treatments are types of 2-stage hepatectomies for removing liver cancer. ALPPS may be more effective than PVO in patients whose disease would traditionally be considered inoperable.

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria: •Patient may have primary or secondary hepatic malignancies with a FLR/TLV < 30% or a FLR/BW ratio of < 0.5 for patients with normal liver function (defined as normal transaminases, normal bilirubin, normal factor V, and normal PT/INR). In case of injury due to chemotherapy, known high grade steatosis, or cholestasis > 50 mmol/L, patient may be enrolled into the trial if FLR/TLV is < 40% or FLR/BW ratio < 0.8.

* Patient must have extensive liver tumors that would require portal vein embolization or a two-stage hepatectomy and portal vein embolization or ligation by the judgment of surgeons in the tumor board.
* Patient may have extrahepatic disease as long as it may be addressed after liver surgery and there is a tumor board decision to proceed with liver resection (mostly applicable to CRC metastases).
* Patient may have received previous chemotherapy.
* In cases of cholestasis, preoperative drainage procedures (PTC or ERCP) are left up to judgement of physicians.
* Patient must be = 18 years of age. The patient population over 65 years old needs to be carefully included based on comorbidities.
* Patient may have undergone previous liver resection.
* Patient's location must be such that proper staging and follow-up may be performed.
* Patient's case must be presented at the Multidisciplinary Meeting attended by hepatobiliary surgeons, oncologists, hepatologists, and radiologists, or must be approved directly by Dr. Strasberg or Dr. Chapman.

Exclusion criteria: •Patient must not have any significant concomitant diseases rendering him/her unsuitable for major liver surgery by the judgment of the physicians involved, especially if the patient is > 65 years old.

* Patient must not have enrolled into a clinical trial within 4 weeks of study entry.
* Patient must not have peritoneal carcinomatosis or other extensive extrahepatic disease.
* Patient must not have advanced stages of carcinoma of the gallbladder (T3/T4)
* Patient must not have issues such as drug and/or alcohol abuse.
* Patient must not need major extrahepatic surgery (e.g. pancreas resection, gastric resection, rectal surgery) within 3 months of study entry.
* Patient must not be a candidate for liver transplantation in case of HCC.
* Patient must not be pregnant or breastfeeding. If a female of childbearing potential, patient must have a negative pregnancy test within 14 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Liver free of tumors [ Time Frame: At 3 months ] [ Designated as safety issue: No ] | 2012 to 2015

SECONDARY OUTCOMES:
rate of hypertrophy over time | 2012 to 2015
Complications of treatment | 2012-2015
Progression of disease | 2012-2015
  Progression free survival
Postoperative liver and renal function | 2012 to 2015

CONTACTS AND LOCATIONS:
Locations (3):
- Washington University, St Louis, Missouri, United States
- Italian Hospital, Department of Surgery, Division of HPB surgery and Liver Transplatn Unit, Buenos Aires, Argentina
- University Hospital Zurich, Division of Visceral and Transplant Surgery, Zurich, Canton of Zurich, Switzerland